CLINICAL TRIAL: NCT04229758
Title: Restarting Anticoagulation After Traumatic Intracranial Hemorrhage (Restart tICrH): a Prospective Randomized Open Label Blinded Endpoint (PROBE) Pragmatic Time-dose, Response Adaptive Clinical Trial
Brief Title: Restarting Anticoagulation After Traumatic Intracranial Hemorrhage
Acronym: Restart tICrH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Truman J Milling Jr, Associate Professor of Neurology, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020090035
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Hemorrhage; Intracranial Hemorrhages; Bleeding; Trauma
Keywords: Anticoagulation; Anticoagulant; Anticoagulants; Restart; Delay; Hemorrhage; ICH; SAH; SDH; DOAC; NOAC; apixaban; rivaroxaban; edoxaban
MeSH Terms: conditions — Hemorrhage; Intracranial Hemorrhages; Wounds and Injuries | interventions — Anticoagulants

STUDY DESIGN:
Intervention Model Description: The trial will employ an innovative adaptive design using time as a dose (1, 2 and 4 weeks) and adapting randomization probabilities to the better performing doses with a PROBE model to minimize surveillance bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 1 week (Experimental): Time to delay the initiation of anticoagulation is determined at randomization. Patients will be randomized to initiate anticoagulation 1 week, 2 weeks, or 4 weeks following injury.
  Interventions: Drug: Anticoagulants
- 2 weeks (Experimental): Time to delay the initiation of anticoagulation is determined at randomization. Patients will be randomized to initiate anticoagulation 1 week, 2 weeks, or 4 weeks following injury.
  Interventions: Drug: Anticoagulants
- 4 weeks (Experimental): Time to delay the initiation of anticoagulation is determined at randomization. Patients will be randomized to initiate anticoagulation 1 week, 2 weeks, or 4 weeks following injury.
  Interventions: Drug: Anticoagulants

INTERVENTIONS:
Drug: Anticoagulants — DOAC for the prevention of thromboembolic events in patients with non-valvular AF or VTE.

SUMMARY:
Primary Objective:

To identify the optimal interval to restart oral anticoagulation after traumatic intracranial hemorrhage that will minimize thrombotic events and major bleeding by performing a response adaptive randomized (RAR) PROBE clinical trial of restarting in anticoagulant-associated traumatic intracranial hemorrhage patients, comparing restart at 1 week to restart at 2 weeks or at 4 weeks, with a primary composite outcome of major thrombotic events and bleeding.

Primary Outcome: 60-day composite of thromboembolic events, defined as DVT, pulmonary emboli, myocardial infarctions, ischemic strokes and systemic emboli, and bleeding events defined as non-CNS major bleeding events (modified BARC3 or above) and worsening index tICrH or new intracranial hemorrhage (ICrH).

Secondary objectives of this trial include:

1. To use the Trauma Quality Improvement Program (TQIP) of the American College of Surgeons - Committee on Trauma (ACS-COT), a well-established and highly respected trauma center oversight mechanism, to translate findings of the trial into practice in a closed loop.
2. To establish a relationship between time of restarting and overall secondary events, i.e. a dose response, that favors early restarting (1 week is better than 2 weeks and 2 weeks is better than 4 weeks.
3. To explore patient centered utility weighting of thrombotic versus bleeding composite endpoint components by: A) 60-day Disability Rating Scale (DRS) 24,25 and modified Rankin Scale (mRS)26; B) Trial patient-reported standard gamble utilities including by race, gender and ethnicity.
4. To explore the composite without DVT in the thrombotic component

DETAILED DESCRIPTION:
Title: Restart tICrH Protocol Synopsis A Prospective Randomized Open Label Blinded Endpoint Response Adaptive Clinical Trial of Timing to Restart Direct Oral Anticoagulants After Traumatic Intracranial Hemorrhage

Objectives: To identify the optimal interval to restart oral anticoagulation after traumatic intracranial hemorrhage that will minimize thrombotic events and major bleeding by performing a response adaptive randomized (RAR) clinical trial of restarting in anticoagulant-associated traumatic intracranial hemorrhage patients, comparing restart at 1 week to restart at 2 weeks or at 4 weeks, with a primary composite outcome of major thrombotic events and bleeding.

Hypotheses: We hypothesize that restarting an oral anticoagulant at one week after anticoagulant-associated traumatic intracranial hemorrhage, compared to delayed restarting, reduces a composite outcome of major thrombotic events and major bleeding.

Study design Prospective, response adaptive randomized, open-label, blinded end-point (PROBE), 40 center national trial Study population -- Approximately 1100 participants with traumatic intracranial hemorrhage and an indication for Direct Oral Anticoagulant Main inclusion criteria

1. Clinician intent to restart a Direct Oral Anticoagulant (DOAC) after anticoagulant-associated traumatic intracranial hemorrhage and equipoise concerning restart of anticoagulation at the specified time intervals.
2. Acute traumatic intracranial hemorrhage on anticoagulation for Atrial Fibrillation (AF) or Venous Thromboembolism (VTE)
3. Patient is higher risk for stroke or other thrombotic events as witnessed by having a CHA2DS2-VASc score of > 3
4. DOAC will be prescribed at label dose with label adjustments for creatinine clearance. DOAC will be at continuation dose, i.e., not initial therapy high doses in the setting of VTE.

Main exclusion criteria

1. Mechanical Valve/Ventricular Assist Device (excludes 1%)
2. SDH >8 mm maximum width or any midline shift at any time point or more than one SDH (excludes 10%)
3. Physician plan to start/restart antiplatelet therapy during trial period (excludes 5%)
4. Abbreviated Injury Scale other than head >3 (excludes 10%)
5. Pregnancy (excludes 0%: median age 81, range 58-99)
6. Inability to understand need for adherence to study protocol
7. Renal function below DOAC label exclusions
8. Any active pathological bleeding (no acute blood most recent CT)
9. Hypersensitivity to drug or other label contraindication
10. Any bleeding that the investigator deems unsafe to restart DOAC at 1 week post injury, or conversely unsafe to hold DOAC to 4 weeks
11. Completion of DOAC therapy expected prior to 60-day primary endpoint, e.g., 3-6-month VTE treatment
12. Concomitant strong inducers/inhibitors of p-gp and CYP3A4
13. Low body weight (<45kg)
14. Inability to swallow

Interventions: • The trial will randomize patients with anticoagulant-associated traumatic intracranial hemorrhage to restart DOAC at 1 week or 2 weeks or 4 weeks, using an adaptive randomization algorithm that increases the probability of patients being randomized to treatment arms with lower event rates.

Primary efficacy outcome: A 60-day composite outcome that includes the following clinical events:

A. Bleeding Events Worsening tICrH/new ICrH

1)Hematoma expansion/new ICrH lesion on imaging 2)causing objective change in clinical status and 3)leading to stop of anticoagulation (must include all three).

Extracranial Major bleeding BARC3a or above definition. B. Thrombotic events Venous Thromboembolism (VTE) It is defined as a clinical diagnosis of acute proximal (popliteal and above) deep vein thrombosis or pulmonary embolus confirmed on imaging (compression ultrasound or venogram for DVT, CT angiography, other angiography or ventilation/perfusion scan for PE) by a radiologist qualified to interpret the scans in a timely manner. If the radiologist cannot or does not attest to acute versus chronic thrombus, the Adjudication Committee will make this determination according to its charter.

Myocardial Infarction (MI) Fourth Universal Definition of Myocardial Infarction.

Stroke New focal neurologic deficit consistent with ischemic stroke and confirmed by a stroke specialist or brain imaging. Brain imaging must be performed but need not be positive if the stroke specialist (neurology, neurosurgery or internal medicine) deems a clinically probable stroke.

Systemic Embolism A clinical diagnosis of extracranial infarction associated with likely thromboembolism and documented by angiography or surgery in the absence of atherosclerotic occlusion.

Cardiovascular death non bleeding Death resulting from an acute myocardial infarction, sudden cardiac death, death due to heart failure, death due to stroke, death due to cardiovascular procedures, and death from other cardiovascular causes 45. A patient who has both this outcome and another thrombotic outcome will only be counted once as this outcome.

Secondary outcomes: Modified Rankin Scale and Disability Rating Scale

Safety outcomes: Incorporated in composite as thrombotic and bleeding events

Statistical analysis: All interim and final analyses will be conducted on the primary outcome, the composite 60-day outcome of thromboembolic events and recurrent hemorrhage. Both thrombotic and bleeding outcomes will be modeled as a function of the three treatment arms in a dose (time)/response (events composite) model. Two Bernoulli models will be used to estimate thromboembolism and recurrent hemorrhage. Each of the rates for the Bernoulli values by dose are θd and δd for thromboembolism and recurrent hemorrhage respectively. These rates are combined to provide a utility function Ud=-θd-δd, so higher values of Ud correspond to the better dose to establish specifically whether at a week is best and generally whether earlier is better than later.

Sample size: 1100

Clinical sites: Approximately 40 trauma center clinical sites in the US.

Recruitment period: Approximately 60 months

Follow-up period: Participants will be followed weekly for 60 days, the study end date.

Special procedures: N/A

Coordinating centers: Seton Dell Medical School Stroke Institute, Coalition for National Trauma Research, Kansas University Medical Center

Sponsor: Seton Dell Medical School Stroke Institute

ELIGIBILITY:
Inclusion Criteria:

Entry into the trial is primarily driven pragmatically by clinician intent to restart a Direct Oral Anticoagulant (DOAC) after anticoagulant-associated traumatic intracranial hemorrhage and equipoise concerning restart of anticoagulation at the specified time intervals. DOAC will be at label dose with label adjustments for creatinine clearance. DOAC will be at continuation dose, i.e. not initial therapy high doses in the setting of VTE.

1. Acute traumatic intracranial hemorrhage on anticoagulation for Atrial Fibrillation (AF) or Venous Thromboembolism (VTE) or both (2,500 patients per year at our 40 sites)
2. Patient is higher risk for stroke or other thrombotic events as witnessed by having a CHA2DS2-VASc score of > 3 (at least 3 of the following risk factors: age greater than 65,( age > 75 counts for two points), history of stroke or TIA, history of heart failure, history of diabetes, history of atherosclerotic vascular disease, female gender, history of hypertension) (Excludes 20% or 500 patients per year)

Exclusion Criteria:

1. Mechanical Valve
2. Ventricular Assist Device (VAD)
3. SDH >8 mm maximum width or any midline shift at any time point or more than one SDH
4. Physician plan to start/restart antiplatelet therapy during trial period
5. Acute Injury Score other than head >=3
6. Pregnancy
7. Inability to understand need for adherence to study protocol
8. Renal function below DOAC label exclusions
9. Any active pathological bleeding (e.g. no acute blood on most recent CT)
10. Hypersensitivity to drug or other label contraindication
11. Any bleeding that the investigator deems unsafe to restart DOAC at 1 week post injury, or conversely unsafe to hold DOAC to 4 weeks
12. Expected completion of DOAC therapy expected prior to 60 day primary outcome, e.g. 3-6 month VTE therapy
13. Concomitant need for strong inducers/inhibitors of p-gp and CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
60 Day Composite of Thrombotic and Bleeding Events | 60 days following index bleeding event
  Composite of Thrombotic events, defined as DVT, PE, MI, Ischemic Strokes, and systemic emboli, cardiovascular death along with bleeding events defined as non-CNS major bleeding, worsening index tICrH, or new intracranial hemorrhage.

SECONDARY OUTCOMES:
60 Day Disability Rating Scale (1-29 with 29 being worse) | 60 days following index bleeding event
  DRS is a scale to measure disability after an injury
60 Day Modified Rankin Scale (1-6 with 6 being worse) | 60 days following index bleeding event
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
Standard Gamble Patient Reported utilities for endpoints | pre-randomization and after endpoints
  Performed prior to randomization and immediately after each endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Truman J Milling, MD, Principal Investigator — Seton Dell Medical School Stroke Institute
Locations (1):
- Dell Seton Medical Center at The University of Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data generated by this project is an essential part of our proposed activities. Following study completion, the DCC staff will follow National Trauma Research Repository (NTRR) and NHLBI's Biologic Specimen and Data Repository Information Coordinating Center (BioLLINCC) policies to upload the study's final de-identified data set, supporting documentation (data dictionary, protocol, consent form, data analysis plans) and any manuscripts. The final data set will be a csv file upload that is consistent with the NTRR data element attributes and characteristics.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of primary manuscript